CLINICAL TRIAL: NCT00946699
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled Study of the Safety and Tolerability of MEDI-551 in Scleroderma
Brief Title: A Study of the Safety and Tolerability of MEDI-551 in Scleroderma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: MI-CP200
Record Dates: First submitted 2009-07-23; First posted 2009-07-27 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Scleroderma
MeSH Terms: conditions — Scleroderma, Diffuse | interventions — inebilizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 1 (Experimental): MEDI-551
  Interventions: Biological: MEDI-551
- 2 (Experimental): MEDI-551
  Interventions: Biological: Placebo
- 3 (Experimental): MEWDI-551
  Interventions: Biological: MEDI-551
- 4 (Experimental): MEDI-551
  Interventions: Biological: MEDI-551
- 5 (Experimental): MEDI-551
  Interventions: Biological: MEDI-551
- 6 (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: MEDI-551 — 0.1 mg/kg
  Arms: 1
Biological: Placebo — 0.3 mg/kg
  Arms: 2
Biological: MEDI-551 — 1.0 mg/kg
  Arms: 3
Biological: MEDI-551 — 3.0 mg/kg
  Arms: 4
Biological: MEDI-551 — 10.0 mg/kg
  Arms: 5
Other: Placebo — Placebo
  Arms: 6

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of intravenously administered MEDI-551 over escalating single doses in adult subjects with Scleroderma

DETAILED DESCRIPTION:
To evaluate the safety and tolerability of escalating single IV doses of MEDI-551 in adult subjects with scleroderma who have at least moderate skin thickening in an area suitable for repeat biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects
* Age ≥ 18 years of age at the time of screening
* Written informed consent and HIPAA authorization (applies to covered entities in the USA only) obtained from the subject/legal representative prior to performing any protocol-related procedures, including screening evaluations
* Must fulfill the American Rheumatism Association (American College of Rheumatology) preliminary classification criteria for systemic sclerosis
* Has at least moderate skin thickening (score of at least 2 by mRTSS) in at least one area suitable for repeat biopsy, such as on the arms, legs, or trunk
* Females of childbearing potential, unless surgically sterile (ie, bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy), has sterile male partner, is at least 2 years post menopause, or practices abstinence, must use 2 effective methods of avoiding pregnancy (including oral, transdermal, or implanted contraceptives, intrauterine device, female condom with spermicide, diaphragm with spermicide, cervical cap, or use of a condom with spermicide by the sexual partner), from screening, and must agree to continue using such precautions through the Early Discontinuation Visit/End of Study (Day 85, single-dose cohorts); cessation of birth control should not occur until 5 half-lives post-cessation of MEDI-551, 5 half-lives is estimated to be 75 days
* Men, unless surgically sterile, must use 2 effective methods of birth control with a female partner and must agree to continue using such contraceptive precautions from Day 1 through the Early Discontinuation Visit/End of Study (Day 85, single-dose cohorts) and for 5 half-lives post-cessation of MEDI-551, 5 half-lives is estimated to be 75 days
* Ability to complete the study period, including follow-up period through Day 85
* Willingness to forego other forms of experimental treatment during the study (Day 1 through the Early Discontinuation Visit/End of Study - Day 85, single-dose cohorts)

Exclusion Criteria:

* History of allergic reactions to any component of the investigational product
* History of coagulation disorders that in the opinion of the investigator would contraindicate skin biopsies
* Has a body weight ≥ 120 kg or < 40 kg
* Has B-cell count in peripheral blood < 50% lower limit of normal (LLN) at screening
* Forced vital capacity (FVC) < 55% predicted, diffusing capacity for carbon monoxide (DLCO) < 40% predicted, pulmonary hypertension requiring treatment with endothelin receptor antagonists or prostacyclin analogues
* Scleroderma renal crisis within the last year, or medically significant malabsorption
* Receipt of any B-cell-depleting biologic therapies at any time, such as rituximab
* Receipt of leflunomide > 20 mg/day within 6 months prior to randomization into the study
* Receipt of the following concomitant medications within 21 days prior to randomization into the study:

  * Prednisone > 30 mg/day or > 0.5 mg/kg
  * Cyclophosphamide
  * Systemic cyclosporine
  * Thalidomide
  * Hydroxychloroquine > 600 mg/day
  * Mycophenolate mofetil > 3 g/day
  * Methotrexate > 25 mg/week
  * Azathioprine > 3 mg/kg/day
  * Concomitant methotrexate and leflunomide
  * Any investigational drug therapy or non-B-cell-depleting biologic therapy (or within 5 half-lives of ingestion, whichever is longer)
* Change in standing daily dosage of the following within 21 days before randomization into the study:

  * Antimalarials
  * Mycophenolate mofetil
  * Methotrexate
  * Leflunomide
  * Azathioprine
  * Systemic corticosteroids
* At screening blood tests (within 21 days prior to randomization into the study), any of the following:

  * Aspartate aminotransferase (AST) > 1.5 × upper limit of the normal range (ULN)unless due to documented myositis
  * Alanine aminotransferase (ALT) > 1.5 × ULN unless due to documented myositis
  * Total bilirubin > ULN, unless because of known Gilbert's disease - Total immunoglobin <500 mg/dl
  * Creatinine > 2.5 mg/dL
  * Neutrophils < 1,500/mm3
  * Platelet count < 75,000/mm3
  * Hemoglobin (Hgb) < 8 g/dL
  * Hemoglobin A1c (HbA1c) > 8% at screening (diabetic subjects only)
  * Positive serum βHCG (pregnancy test)
* Lactating woman
* Herpes zoster infection within 3 months before randomization
* A history of severe viral infection as judged by the investigator, including severe infections of either cytomegalovirus or the herpes family such as disseminated herpes, herpes encephalitis, ophthalmic herpes
* At screening, positive tests for active hepatitis A, hepatitis B surface antigen (HbsAg), Hepatitis B core antibody (HbcAb) or hepatitis C serology, or human immunodeficiency virus-1 or -2 (HIV-1/2). False positive tests are not included.
* Deep space/tissue infection (eg, fasciitis, abscess, osteomyelitis, or infected joint replacements) within 1 year before randomization into the study
* Any opportunistic infection or serious infection (in the opinion of the investigator) within 6 months prior to screening
* Any of the following within 21 days before randomization into the study:

  * Clinically significant active infection, including ongoing, chronic infection
  * Any infection requiring hospitalization or treatment with IV anti-infectives
* Completion of a course of oral anti-infectives within 14 days before randomization into the study
* Any acute illness or evidence of clinically significant active infection, such as fever ≥ 38.0 degrees C (≥ 100.5 degrees F) at screening or at Day 1
* Evidence of active tuberculosis (TB), either treated or untreated, or latent TB without completion of an appropriate course of treatment or appropriate ongoing prophylactic treatment. Evaluation and treatment will be according to the local standard of care and may consist of history and physical examinations, and/or chest X ray, and/or TB test (eg. purified protein derivative) testing, with the standard of care as determined by local guidelines
* History of primary immunodeficiency or underlying condition that predisposes the subject to infection (eg, splenectomy)
* Receipt of any live or attenuated vaccine within 21 days before randomization into the study or anticipated to be given within 5 half-lives of the last dose of investigational product administration, half-life is estimated to be approximately 15 days. Therefore, receipt of live attenuated vaccine should be avoided for 75 days post dose of investigational product
* Medically indicated adult immunizations that are not current (eg, pneumococcal vaccine)
* Current evidence of alcohol, drug or chemical abuse, or a recent history of such abuse < 1 year prior to randomization into the study
* History of cancer except basal cell carcinoma treated with apparent success with curative therapy ≥ 1 year prior to randomization into the study
* Major surgery within 8 weeks before randomization into the study or elective surgery planned from screening through the Early Discontinuation Visit/End of Study (Day 85, single-dose cohorts)
* History of any disease, evidence of any current disease (other than scleroderma), any finding upon physical examination, chest x-ray, or any laboratory abnormality that, in the opinion of the investigator or medical monitor, may compromise the safety of the subject in the study or confound the analysis of the study
* Any institutionalized individual
* Employees of the clinical study site or any other individuals involved with the conduct of the study, or immediate family members of such individuals
* Concurrent enrollment in another clinical study with the exception of observational or interventional studies that do not involve therapeutic strategies or invasive diagnostic tests
* Concurrent enrollment in another clinical study with an investigational product administered within 4 weeks prior to Day 1 or within 5 half-lives of the investigational product, whichever is longer
* Known sensitivity to acetaminophen/paracetamol, diphenhydramine, and methylprednisolone or equivalent glucocorticoid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-03; Primary Completion 2012-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
The safety and tolerability of MEDI-551 will be assessed primarily by summarizing treatment-emergent AEs and SAEs. | Day 85

SECONDARY OUTCOMES:
The secondary endpoints of the study are to assess the PK, IM, and PD of single IV doses of MEDI-551 in adult subjects with scleroderma. Pharmacodynamics will be assessed by numbers of B cells in blood and skin. | Day 85

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — MedImmune LLC
Locations (14):
- United States (12):
  - Research Site, Loma Linda, California
  - Research Site, Redwood City, California
  - Research Site, Farmington, Connecticut
  - Research Site, Shreveport, Louisiana
  - Research Site, Worcester, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, New Brunswick, New Jersey
  - Research Site, Great Neck, New York
  - Research Site, Durham, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Dallas, Texas
- Research Site, Winnipeg, Manitoba, Canada
- Research Site, London, United Kingdom

REFERENCES:
- [Derived] Schiopu E, Chatterjee S, Hsu V, Flor A, Cimbora D, Patra K, Yao W, Li J, Streicher K, McKeever K, White B, Katz E, Drappa J, Sweeny S, Herbst R. Safety and tolerability of an anti-CD19 monoclonal antibody, MEDI-551, in subjects with systemic sclerosis: a phase I, randomized, placebo-controlled, escalating single-dose study. Arthritis Res Ther. 2016 Jun 7;18(1):131. doi: 10.1186/s13075-016-1021-2. PMID 27267753